CLINICAL TRIAL: NCT03470753
Title: The Impact of Home Exercise Program Delivery Type on Exercise Compliance and Clinical Outcomes for Musculoskeletal Pain
Brief Title: Impact of Home Exercise Delivery on Compliance & Outcomes for Musculoskeletal Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dan Rhon (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Dan Rhon, Researcher, Brooke Army Medical Center
Organization: Brooke Army Medical Center (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C.2017.093d
Record Dates: First submitted 2018-02-07; First posted 2018-03-20 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Chronic Pain; Compliance, Patient; Chronic Low Back Pain; Knee Pain Chronic
MeSH Terms: conditions — Chronic Pain; Patient Compliance

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Exercise Amount (Active Comparator): Phase 1: 2 or 4 exercises.
  Interventions: Other: Number of Exercises; Other: Type of Instruction
- Type of instruction (Active Comparator): Phase 1: Handout on paper versus handout and visual demonstration/performance.
  Interventions: Other: Number of Exercises; Other: Type of Instruction
- Delivery Type (Active Comparator): Phase 2: Handout vs electronic delivery
  Interventions: Other: Delivery Type; Other: Mobile Reminder
- Reminder Type (Experimental): Phase 2: Mobile reminders vs no mobile reminders
  Interventions: Other: Delivery Type; Other: Mobile Reminder

INTERVENTIONS:
Other: Number of Exercises — Subjects will receive either 2 or 4 exercises to evaluate the short-term recall and performance.
  Arms: Exercise Amount; Type of instruction
Other: Type of Instruction — The type of instruction in phase 1 will be compared: Instruction by providing a handout only vs being instructed by a provider and practiced by the patient with provider feedback.
  Arms: Exercise Amount; Type of instruction
Other: Delivery Type — In phase 2 subjects will be provided 4 exercises using only a handout vs delivered to them electronically with the addition of a video.
  Arms: Delivery Type; Reminder Type
Other: Mobile Reminder — A text-message based mobile reminder tool will be utilized to engage with subjects via texting on a daily basis to provide reminders and encouragement to perform their home exercises.
  Arms: Delivery Type; Reminder Type

SUMMARY:
Patients seeking care for chronic low back or knee pain will be recruited for enrollment, and randomized within two phases (retention and compliance). Patients will consent to a 2-step study design, with independent randomization for each. The initial step will assess retention based on 4 different exercise prescription strategies. This will be assessed short-term, and then the 2nd step will consist of a second independent randomization to receive different reminder strategies to determine their influence on exercise compliance at home.

DETAILED DESCRIPTION:
Patients seeking care for their chronic low back or knee pain will be recruited to participate in a trial investigating the value of different exercise and education prescription strategies as well as strategies to determine the influence of various exercise reminder strategies. On day 1 of enrollment, patients will be randomized and instructed in two different types and amounts of exercises, as well as two types of delivery strategies. The ability to recall and perform these exercises will be assessed 20 minutes after completion of the instructional period (retention). In phase 2, patients will be randomized to receive different reminder strategies (none, email, text, and/or video) and their compliance assessed over a 1 month period (compliance). Self-reported compliance over the first month, and health care utilization outcomes will be analyzed for the 1 year following completion of the 1 month period, in all groups.

ELIGIBILITY:
Inclusion Criteria:

1. The primary complaint of low back pain or knee pain and is not actively seeking care for their contralateral knee.
2. The current episode for the injury is 6 weeks or greater
3. A home exercise program is appropriate as part of the management plan for their injury on the first day
4. Between the age of 18 and 65 years.
5. Own and utilize a smart phone
6. Read and speak English well enough to interact with the smart phone-based tool.
7. Able and willing to come in for follow-up at 1-month.

Exclusion Criteria:

1. History of prior surgery to the lower extremities or spine
2. Already receiving or have received treatment for this episode of pain within the past 6 months.
3. Medical "red flags" of a potentially serious condition including cauda equina syndrome, major or rapidly progressing neurological deficit, fracture, malignancy, joint infection, or systemic disease
4. If participating with low back pain, known current pregnancy or history of pregnancy in the last 6 months
5. Exiting military health system in the next 2 months, pending litigation, or pending a medical separation board.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2018-01-12 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
Performance Assessment Tool | 1-month
  A locally developed tool designed to meet the needs of assessing both exercise retention and compliance. It will capture the subject's ability to recall the name of an exercise, the prescribed sets and repetitions, and the ability to perform an exercise using a 4-point ordinal scale
Compliance | 1-month
  Subjects will be asked to submit self-reported daily compliance logs.

SECONDARY OUTCOMES:
Patient Reported Outcomes Measurement Information Systems (PROMIS) 57 (v2.0) | 1-month
  The PROMIS 57-item short form efficiently assesses several outcomes important to patients with chronic low back and knee pain including pain intensity and interference, sleep disturbance, anxiety, depression, fatigue, and social role participation using items developed with rigorous methodology and patient input.
Patient Acceptable Symptom State (PASS) | 1-month
  the PASS as a global, dichotomized single-item score indicating if patients are satisfied with the current state of their symptoms.
Self-perception on Physical Health and Ability to Return to Work or Full Duty | 1-month
  This survey consists of a total of 9 questions, 5 of them modified from the Short Form-36. It asks questions related to the subject's perception of their physical health. The first 5 questions are related to the subject's perception of ability to return to work or full duty, the need for additional healthcare for their current condition, and function at the level that they feel is expected of them. The final 4 questions ask about their perception of general physical health.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Rhon, DSc, Principal Investigator — Brooke Army Medical Center
Locations (1):
- Brooke Army Medical Center, San Antonio, Texas, United States

REFERENCES:
- [Background] Jordan JL, Holden MA, Mason EE, Foster NE. Interventions to improve adherence to exercise for chronic musculoskeletal pain in adults. Cochrane Database Syst Rev. 2010 Jan 20;2010(1):CD005956. doi: 10.1002/14651858.CD005956.pub2. PMID 20091582
- [Background] Bollen JC, Dean SG, Siegert RJ, Howe TE, Goodwin VA. A systematic review of measures of self-reported adherence to unsupervised home-based rehabilitation exercise programmes, and their psychometric properties. BMJ Open. 2014 Jun 27;4(6):e005044. doi: 10.1136/bmjopen-2014-005044. PMID 24972606
- [Background] Chou R, Huffman LH; American Pain Society; American College of Physicians. Nonpharmacologic therapies for acute and chronic low back pain: a review of the evidence for an American Pain Society/American College of Physicians clinical practice guideline. Ann Intern Med. 2007 Oct 2;147(7):492-504. doi: 10.7326/0003-4819-147-7-200710020-00007. PMID 17909210
- [Background] Hayden JA, van Tulder MW, Tomlinson G. Systematic review: strategies for using exercise therapy to improve outcomes in chronic low back pain. Ann Intern Med. 2005 May 3;142(9):776-85. doi: 10.7326/0003-4819-142-9-200505030-00014. PMID 15867410
- [Background] Jack K, McLean SM, Moffett JK, Gardiner E. Barriers to treatment adherence in physiotherapy outpatient clinics: a systematic review. Man Ther. 2010 Jun;15(3):220-8. doi: 10.1016/j.math.2009.12.004. Epub 2010 Feb 16. PMID 20163979
- [Background] Holcomb LS. A Taxonomic Integrative Review of Short Message Service (SMS) Methodology: A Framework for Improved Diabetic Outcomes. J Diabetes Sci Technol. 2015 Apr 30;9(6):1321-6. doi: 10.1177/1932296815585132. PMID 25934517